CLINICAL TRIAL: NCT01978223
Title: Case-control Study to Evaluate the Vaccine Effectiveness of RotarixTM Against Rotavirus Severe Gastroenteritis Among Hospitalised Children Aged 12 Weeks to < 5 Years, in Venezuela
Brief Title: Effectiveness of RotarixTM Vaccine in Children Aged Between 12 Weeks to < 5 Years, Hospitalised for Severe Gastroenteritis
Status: Withdrawn | Type: Observational
Why Stopped: As vaccine coverage rates have drastically improved in Venezuela, the study lost its objective to show positive impact of the vaccine to stimulate higher usage
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116494
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Infections, Rotavirus
Keywords: Rotarix™; Case-control; Venezuela; Vaccine effectiveness; Rotavirus Severe Gastroenteritis; Children; Hospitalised
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample

GROUPS / COHORTS (2):
- Cases: Children hospitalised for SGE, aged 12 weeks to < 5 years at the time of hospital admission/ED stay and whose stool samples test positive for RV by enzyme linked immunosorbent assay (ELISA) at a GSK designated laboratory.
  Interventions: Procedure: Stool sample collection
- Controls: Children hospitalised for SGE, aged 12 weeks to < 5 years at the time of hospital admission/ ED stay, whose stool samples test negative for RV by enzyme linked immunosorbent assay at a GSK designated laboratory and who will be matched to the cases by date of birth and the hospital of admission/ ED stay.
  Interventions: Procedure: Stool sample collection

INTERVENTIONS:
Procedure: Stool sample collection — Stool samples will be collected from all children enrolled in the study, within 48 hours of admission to the hospital/ ED. Stool samples will be tested to determine the presence or absence of rotavirus (RV). Additionally, for RV-positive cases, the stool samples will be tested to determine the RV genotypes.

SUMMARY:
This study aims to estimate the effectiveness of Rotarix™ vaccine against Rotavirus severe gastroenteritis (RV SGE) among hospitalised children aged between 12 weeks and < 5 years, in Venezuela and to assess the current disease burden after introduction of the vaccine.

DETAILED DESCRIPTION:
The data generated in this study will be useful for public health officers and policy makers in confirming the country-wide public health benefit of Rotarix™.

No vaccine will be administered during this study.

ELIGIBILITY:
Inclusion Criteria:

For SGE subjects:

* A male or female child aged 12 weeks to < 5 years at the time of hospital admission/ ED stay. The subject becomes ineligible on the fifth birthday.
* Subject admitted to (or who will have an ED stay at) the study hospital(s) for SGE during the study period.
* Onset of SGE ≤ 14 days prior to admission/ ED stay.
* Written/thumb printed informed consent obtained from the parent(s)/legally acceptable representative(s) (LAR (s)) of the subject.

For Cases:

• Laboratory confirmed (i.e. by ELISA) RV-positive stool sample collected at hospital admission/ ED stay or during the first 48 hours of hospitalisation.

For Controls:

* Subject admitted to (or who will have an ED stay at) the same study hospital(s) for SGE as that of the case during the study period.
* Laboratory confirmed (i.e. by ELISA) RV-negative stool sample collected at hospital admission/ ED stay or during the first 48 hours of hospitalisation.
* Subjects born within ± 2 weeks from the date of birth of the case.

Exclusion Criteria:

For SGE subjects:

* Child in care.
* Hospitalisation is unrelated to GE.
* Onset of SGE > 48 hours after admission to (or ED stay at) the hospital.
* Subject has digestive tube anomalies, chronic gastrointestinal disease or uncorrected congenital abnormalities.
* Subject with immunodeficiency.
* Subjects who live out of the federative entity where hospital(s) are located.

For Controls:

• Subject has previously participated as case in this study.

Ages: 12 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 12 weeks to < 5 years, hospitalised for SGE in the study hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Full vaccination status of Rotarix™ (2 doses) with the vaccine administered at least 2 weeks before hospitalisation in RV-positive SGE children (cases) compared to RV-negative SGE children (controls). | During hospitalisation and after discharge (approximately 12 months from study initiation).

SECONDARY OUTCOMES:
Full/partial vaccination status (at least one dose of Rotarix™) with the vaccine administered at least 2 weeks before hospitalisation in RV-positive SGE children (cases) compared to RV-negative SGE children (controls). | During hospitalisation and after discharge (approximately 12 months from study initiation).
Occurrence of specific RV genotype among the enrolled RV SGE children with full/partial vaccination status (at least one dose of Rotarix™ with the vaccine is administered at least 2 weeks before hospitalisation). | During hospitalisation and after discharge (approximately 12 months from study initiation).
Occurrence of RV SGE in children by age at hospitalisation with full/partial vaccination status (at least one dose of Rotarix™ with the vaccine administered at least 2 weeks before hospitalisation). | During hospitalisation and after discharge (approximately 12 months from study initiation).
Occurrence of RV SGE in children by severity with assessment of severity of RV SGE cases by the Vesikari scale. | During hospitalisation and after discharge (approximately 12 months from study initiation).
Occurrence of SGE [≤14 days prior to admission/ Emergency Department (ED) stay] among all hospitalised children. | During hospitalisation and after discharge (approximately 12 months from study initiation).
Occurrence of RV SGE hospital admissions/ ED stays among children hospitalised at the study hospital(s) for SGE. | At hospital admission/ ED stay or during the first 48 hours of hospitalisation.
Occurrence of RV SGE admissions/ ED stays by age of the child (at hospitalisation) and month of year. | During hospitalisation and after discharge (approximately 12 months from study initiation).
Occurrence of RV genotypes among children admitted to (or who have had an ED stay at) the study hospital(s) for SGE. | During hospitalisation and after discharge (approximately 12 months from study initiation).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline